CLINICAL TRIAL: NCT07379021
Title: The Effect of Mindfulness-Based Emotion Regulation Training on Fear and Emotion Regulation in Hospitalized Children
Brief Title: Mindfulness-Based Emotion Regulation Training for Hospitalized Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 30.2.ATA.0.01.00
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Fear; Child, Only; Hospitalism in Children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training (Experimental): In addition to routine nursing care, children in the intervention group will receive the 'Mindfulness-Based Emotion Regulation Training Programme' developed by the researcher.
  * T1 (Pre-test): On the first day of admission, the scales will be administered before the first training session.
  * Application: For 5 consecutive days, once a day, structured sessions (breathing exercises, emotion recognition, body scan, etc.), each lasting approximately 20 minutes, will be conducted in the child's own room with tablet/visual material support and under the guidance of a researcher. During the application, the quietness of the environment and the child's attention will be maintained in a standard manner.
  * T2 (Post Test): At the end of the 5th day (after the final session), the scales will be re-administered to evaluate the programme's effectiveness. Completing the forms will take an average of 15-20 minutes.
  Interventions: Behavioral: training
- control (No Intervention): Children in the control group will not receive any mindfulness training from the researcher; only the clinic's routine nursing care and treatment procedures will be applied.
  * T1 (Pre-test): Scales will be administered on the first day of admission, prior to routine care.
  * T2 (Post-Test): Scales will be administered again on the 5th day of hospitalisation to complete data collection. Completing the forms will take an average of 15-20 minutes.

INTERVENTIONS:
Behavioral: training — In addition to routine nursing care, children in the intervention group will receive the 'Mindfulness-Based Emotion Regulation Training Programme' developed by the researcher.
  Arms: training

SUMMARY:
Hospitalization and medical procedures are a significant source of stress and anxiety for school-age children aged 7-11, who, due to their cognitive development, can perceive events but lack the capacity to cope effectively. The main objective of this project is to examine the effect of Mindfulness-Based Emotion Regulation Training, which will be applied to children aged 7-11 hospitalized in the pediatric clinic, on developing children's emotion regulation skills and reducing their fear levels related to the hospital. The research is a randomized controlled trial to be conducted between April 2026 and April 2027. Data will be collected using the "Child and Parent Introduction Form," the "Emotion Regulation Scale for Children and Adolescents," and the "Medical Procedure Fear Scale." While distraction techniques frequently used in the literature offer a quick and effective solution at the time of the procedure, this project differs in that it aims to provide children with sustainable emotion regulation skills that they can use not only at that moment but also in later stages of the illness and in future life events. As a result of the project, it is expected that the implemented training will increase adaptive emotion regulation strategies in children, significantly reduce medical fear and anxiety, and provide an evidence-based nursing intervention that will facilitate children's compliance with treatment.

DETAILED DESCRIPTION:
The main objective of this project is to examine the effect of Mindfulness-Based Emotion Regulation Training, which will be applied to children aged 7-11 hospitalized in the pediatric clinic, on developing children's emotion regulation skills and reducing their fear levels related to the hospital. The research is a randomized controlled trial to be conducted between April 2026 and April 2027. Data will be collected using the "Child and Parent Introduction Form," the "Emotion Regulation Scale for Children and Adolescents," and the "Medical Procedure Fear Scale." While distraction techniques frequently used in the literature offer a quick and effective solution at the time of the procedure, this project differs in that it aims to provide children with sustainable emotion regulation skills that they can use not only at that moment but also in later stages of the illness and in future life events. As a result of the project, it is expected that the implemented training will increase adaptive emotion regulation strategies in children, significantly reduce medical fear and anxiety, and provide an evidence-based nursing intervention that will facilitate children's compliance with treatment.

Control Group: Children in the control group will not receive any mindfulness training from the researcher; only the clinic's routine nursing care and treatment procedures will be applied.

* T1 (Pre-test): Scales will be administered on the first day of admission, prior to routine care.
* T2 (Post-Test): Scales will be administered again on the 5th day of hospitalisation to complete data collection. Completing the forms will take an average of 15-20 minutes.

Intervention Group: Children in the intervention group will receive the 'Mindfulness-Based Emotion Regulation Training Programme' developed by the researcher in addition to routine nursing care.

* T1 (Pre-test): Scales will be administered on the first day of admission, before the first training session.
* Application: For 5 consecutive days, once a day, structured sessions (breathing exercises, emotion recognition, body scan, etc.), each lasting approximately 20 minutes, will be conducted in the child's own room with tablet/visual material support and under the guidance of the researcher. During the application, the quietness of the environment and the child's attention will be maintained in a standard manner.
* T2 (Post Test): At the end of the 5th day (after the final session), the scales will be re-administered to evaluate the programme's effectiveness. Completing the forms will take an average of 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 7 and 11 years old,
* Have a planned hospital stay of at least four days,
* Be able to speak and understand Turkish,
* Be able to read and write (to complete questionnaires),
* The child and parent must be willing to participate in the study.

Exclusion Criteria:

* The child has a hearing/speech problem that prevents them from communicating,
* The child has severe pain or acute respiratory distress that prevents them from participating,
* The child has a known psychiatric diagnosis,
* The child has previously received similar mindfulness training

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Scale for Children and Adolescents: | 1 year
  The scale was adapted by Gullone and Taffe (2012) from the Emotion Regulation Scale developed by Gross and John (2003) for an adult sample. The scale was adapted into Turkish by Tetik and Önder in 2021. The scale is a self-assessment tool designed to evaluate differences in the use of two emotion regulation strategies. The scale includes statements such as 'I control my emotions by not showing them.' The scale consists of 'two subscales, reappraisal and suppression, and 10 items.' The assessment is conducted using a 5-point Likert-type rating scale. Items 1, 3, 5, 7, 8, and 10 represent the reappraisal subscale, while items 2, 4, 6, and 9 represent the suppression subscale. High scores on the subscales indicate frequent use of the emotion regulation strategy represented by that subscale. The Cronbach's alpha internal consistency coefficient ranged from .82 to .86 for the reappraisal subscale and from .69 to .79 for the suppression subscale.
Medical Procedure Fear Scale | 1 year
  Developed by Marion Bloom et al. in 1985, this scale measures children's fears related to medical procedures and treatments. The validity and reliability study of the scale in Turkey was conducted by Alak (1993). The scale contains items such as 'I am afraid the doctor will hurt me' and 'I am afraid of going to the hospital' and is a 3-point Likert scale (0 = Never, 1 = Sometimes, 2 = Very much). Medical fears are addressed in 29 questions. The scale consists of four sub-dimensions. The Cronbach's alpha for the scale was found to be 0.93. The minimum score obtainable from the scale is 29, and the maximum score is 87. An increase in score indicates an increase in medical fear.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.